CLINICAL TRIAL: NCT02133989
Title: Ticlopidine+Ginkgo Biloba Versus Clopidogrel in Clopidogrel Resistant Patients Undergoing Cartoid Artery Stent Placement
Brief Title: Clopidogrel Resistance and Embolism in Carotid Artery Stenting
Acronym: CRECAS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Yuyu Pharma, Inc. (Industry)
Responsible Party: Principal Investigator, Oh Young Bang, MD, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-06-123
Record Dates: First submitted 2014-04-28; First posted 2014-05-08 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Carotid Stenosis
Keywords: Carotid stenosis; Stenting; Clopidogrel resistance; Stroke, ischemic
MeSH Terms: conditions — Carotid Stenosis; Ischemic Stroke | interventions — Ticlopidine; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ticlopidine+Ginko biloba (Experimental): Switch to ticlopidine + ginko biloba
  Interventions: Drug: Ticlopidine + Ginko biloba
- Clopidogrel (Active Comparator): Keep clopidogrel
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticlopidine + Ginko biloba — ticlopidine hydrochloride 250mg, ginko leaf ext. 80mg, twice daily
  Other Names: Yuclid
  Arms: Ticlopidine+Ginko biloba
Drug: Clopidogrel — clopidogrel bisulfate 97.875mg(75mg as clopidogrel)
  Other Names: Plavix
  Arms: Clopidogrel

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of the ticlopidine + ginko biloba compared to clopidogrel in clopidogrel resistant patients undergoing carotid artery stent placement. The investigators hypothesized that ticlopidine + ginko biloba is superior than clopidogrel in terms of post-stent ischemic lesions in these patients without serious complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for stent implantation due to carotid stenosis
* Patients resistant to clopidogrel defined by platelet inhibition rate <20% measured by Verify Now before carotid stenting
* Patients with informed consent

Exclusion Criteria:

* Antiplatelet therapy other than aspirin, clopidogrel, or ticlopidine
* Unable to perform MRI scans
* Patients with hematologic abnormalities including neutrophil <1500/ul, platelet <100,000/uL, or AST/ALT >120 U/L
* Unsuitable for participation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2014-06; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
New ischemic lesion on diffusion-weighted imaging (DWI) | within 24 hours after carotid stenting
  Presence of new ischemic lesion in the ipsilesioinal hemisphere on DWI after carotid stening

SECONDARY OUTCOMES:
Number and Volume of new ischemic lesions on DWI | within 24 hours after carotid stenting
Benign and malignant microembolic signals (MES) on transcranial Doppler (TCD) | within 24 hours after carotid stenting
Ischemic stroke or transient ischemic attack (TIA) | within 30 days after carotid stenting
Change of clopidogrel resistance | 1 day after carotid stenting
  Change of clopidogrel resistance measured by Verify now (P2Y12)
Pucture site hematoma | within 30 days after carotid stenting
Mycocardial infarction | within 30 days after carotid stenting
Death | within 30 days after carotid stenting
Hematological abnormalities | within 30 days after carotid stenting
  Neutrophil <1500/uL Platelet <100,000/uL AST or ALT >120 U/L

CONTACTS AND LOCATIONS:
Overall Officials: Oh Young Bang, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Oh Young Bang, Seoul, South Korea

REFERENCES:
- [Derived] Chung JW, Kim SJ, Hwang J, Lee MJ, Lee J, Lee KY, Park MS, Sung SM, Kim KH, Jeon P, Bang OY. Comparison of Clopidogrel and Ticlopidine/Ginkgo Biloba in Patients With Clopidogrel Resistance and Carotid Stenting. Front Neurol. 2019 Jan 30;10:44. doi: 10.3389/fneur.2019.00044. eCollection 2019. PMID 30761076